CLINICAL TRIAL: NCT02116595
Title: Alterations in Urine pH With Differing Diet Net Acid Loads
Brief Title: Urine pH and Diet Net Acid Load
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not funded
Sponsor: University of California, San Francisco (Other)
Collaborators: optimal wellness labs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: UPH&DNAE
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- feeding a high acid diet x 24 hrs (Experimental): 2 diets, one low and one high net acid loads
  Interventions: Other: high or low acid diet
- low acid diet (Active Comparator)
  Interventions: Other: high or low acid diet

INTERVENTIONS:
Other: high or low acid diet — high or low acid diets

SUMMARY:
Presently, the gold standard for testing diet acid intake is a urine collection done for many hours, usually 24 hours, which must be analyzed in a research lab for "net acid excretion". So, getting information about diet acid intake is difficult. Many people have suggested doing a much simpler test, which is checking the pH of the urine when you wake up. But, no one has studied if this simpler method is a valid method for estimating the 24 hour net acid excretion. Diet acid load may be important in many diseases associated with aging, such as loss of bone and muscle, and the development of kidney disease.

DETAILED DESCRIPTION:
the primary outcome variable is morning urine pH and 24 hour urine net acid excretion

ELIGIBILITY:
Inclusion Criteria:

* no medical or psychological problems
* able to come to UCSF for study

Exclusion Criteria:

* pregnant or trying to become pregnant
* Hg < 10
* abnormal screening labs
* anyone unable to follow study directions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
high acid diet | 6 months
  correlation between first morning urine pH and 24 hour net acid excretion
low acid diet | 6 months
  correlation between first morning urine pH and 24 hour net acid excretion

CONTACTS AND LOCATIONS:
Overall Officials: lynda frassetto, md, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States